CLINICAL TRIAL: NCT02473601
Title: To Observe Mivacurium Chloramine Muscle Relaxation Effect in the Operation Anesthesia Patients With Liver Cirrhosis
Brief Title: Mivacurium Chloramine Muscle Relaxation Effect in Patients With Liver Cirrhosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Collaborators: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, zhaoxiaoyong, Anesthesiologist, Tang-Du Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015001
Record Dates: First submitted 2015-05-24; First posted 2015-06-16 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Liver Dysfunction
Keywords: mivacurium chloramine; patients with liver cirrhosis; muscle relaxation effect
MeSH Terms: conditions — Liver Diseases | interventions — Mivacurium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mivacurium Chloride by liver dysfunction (Experimental): Mivacurium Chloride 0.2mg/kg,during anesthesia induction. Mivacurium Chloride 6mg/kg/h,during anesthesia maintenance
  Interventions: Drug: Mivacurium Chloride
- Mivacurium Chloride by normal liver function (Other): Mivacurium Chloride 0.2mg/kg,during anesthesia induction. Mivacurium Chloride 6mg/kg/h,during anesthesia maintenance
  Interventions: Drug: Mivacurium Chloride

INTERVENTIONS:
Drug: Mivacurium Chloride — Anesthesia induction:
  Intravenous injection of midazolam 0.05 mg/kg,Etomidate 0.3 mg/kg,Sufentanil 0.5 g/kg,TOF detection and adjustment of the first twitch height (T1)100%, Mivacurium Chloramine 0.07 mg/kg intraveous injecting in 5 minutes.
  Anesthesia maintenance:
  Two groups of sevoflurance 1%~8% inhalation anesthesia plus intravenous infusion of remifentanil 0.05～0.2 µg/kg/min,Mivacurium Chloramine 6mg/kg/h, Appropriate supplementary analgesia dose of sufentanil before skin incision and the abdomen was closed. The two groups were maintained until the Bis value was 40 ~ 60. PetCO2 was 30 ~ 35mmHg. Hemodynamic fluctuations did not exceed 20% of the baseline value.At least 20 minutes before the operation stopping Mivacurium infusion,Before the end of operation 5-10 minutes stopping infusion of remifentanil and sevoflurane.
  Other Names: mivacurium; mivacron

SUMMARY:
Observed the muscle relaxation of mivacurium in patients with liver cirrhosis.Clear of mivacurium in patients with liver cirrhosis without muscle relaxant accumulation and delayed recovery phenomenon

DETAILED DESCRIPTION:
The liver is an important organ of the body to maintain life activities, material and energy metabolism, and the main organ of biotransformation and elimination of toxic substances and drugs, have many complex functions. Anesthetic drugs mostly through liver transformation and degradation.Liver cirrhosis, liver cancer patients due to abnormal liver dysfunction and liver metabolism, Most of the muscle relaxant prone to muscle relaxant accumulation and delayed recovery of patients with liver cirrhosis.

Mivacurium is a new type of non depolarizing muscle relaxants，has the characteristics of rapid onset, short duration of action. Mivacurium can produce similar clinical effect of depolarizing muscle relaxant succinylcholine, and rapidly be blood Che catabolism, Without liver metabolism. It can either as a single vein for medicinal endotracheal intubation, or as maintain continuous intravenous auxiliary anesthesia drug , is a muscle relaxant to shorten the clinical anesthesia recovery period ideal.

ELIGIBILITY:
Inclusion Criteria:

* Patients volunteered for the clinical research and signed a written informed consent
* Experimental group patients is cirrhosis of the liver (liver function grade Child - Pugh, grade A) ready to abdominal surgery patients; The control group was no cirrhosis, ready to abdominal surgery patients
* Aged 18 ~ 60
* BMI<28kg/㎡
* The American society of anesthesiologists (ASA) class I ~ II

Exclusion Criteria:

* Systolic blood pressure ≥180 mm Hg or < 90 mm Hg, diastolic blood pressure ≥110 mm Hg or < 60 mm Hg
* Serious heart, brain, liver, kidney, lung, endocrine diseases or serious infection
* Patients with difficult airway (such as Mallampati airway class III, airway abnormalities, etc.)
* HR < 50 times/min
* The patient had a history of mental illness or chronic psychiatric drugs, chronic pain medication history
* History of alcoholism
* Patients with neuromuscular system disease
* Has a tendency to malignant hyperthermia
* The patient used to test drug allergies or other contraindications
* Over the past 30 days participated in other clinical drug research

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
TOF ratio | Time from administration to TOF (T4/T1) values recovered to 90%,an expected average of 25-30 minutes

SECONDARY OUTCOMES:
Steward score | Time from the end of operation to extubation period,an expected average of 15 minutes
Ramsay score | Time from the end of operation to extubation period,an expected average of 15 minutes
Mivacurium induced time | Time from intravenous injection of mivacurium to T1 reached the maximum inhibition time,an expected average of 3-5 minutes
Clinical duration of action | Time from the Mivacurium injection up to recovery from the neuromuscular blockade to 25% of the initial value, an expected average of 12-20 minutes
Total duration of action | Time from the Mivacurium injection up to recovery from the neuromuscular blockade to 95% of the initial value,an expected average of 25-30 minutes
Recovery index | Time between a 25% and 75% recovery from a neuromuscular blockade,an expected average of 6-8 minutes
Change of the mean arterial pressure (MAP) and heart rate (HR) during pulling out the endotracheal tube period | 10 minutes before pulling the endotracheal tube, the moment of pulling the endotracheal tube immediately, pull out the endotracheal tube after 5 min

CONTACTS AND LOCATIONS:
Overall Officials: zhao xiaoyong, master, Principal Investigator — Shanxi Province, Xi'an city Baqiao District Temple Road, No. 1 Tangdu Hospital; sun meiyan, master, Principal Investigator — Shanxi Province, Xi'an city Baqiao District Temple Road, No. 1 Tangdu Hospital
Locations (1):
- Tangdu hospital, Xi’an, Shanxi, China